CLINICAL TRIAL: NCT04751019
Title: The Use of Amber Glasses in Improving Sleep and Reducing the Use of Hypnotic Medication in an Inpatient Mental Health Setting: Pilot Study
Brief Title: The Use of Amber Glasses in Improving Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Surrey and Borders Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 262339
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Sleep Disturbance; Insomnia
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Amber Glasses — It is hoped that the use of amber glasses to complement the natural sleep-wake by inducing a perceived 'physiological darkness' to aid the secretion of melatonin should help sleep and reduce the use of hypnotic medication

SUMMARY:
The use of amber glasses will aid the patient to fall asleep without the need for the use of hypnotic medication.

DETAILED DESCRIPTION:
Sleep disturbance and insomnia is extremely common and affects up to 30% of adults at any given time. Moreover, sleep disturbance is known to be particularly prevalent in patients suffering from mental illness including affective disorders, schizophrenia, anxiety (Baglioni, 2016). We hypothesise that the use of amber glasses will aid the time taken to fall asleep without the need for the use of hypnotic medication.A prospective study looking at 15 new patients admitted to one mental health ward will be undertaken. Data will be collected on twice weekly basis on the patient's use of: amber glasses alone, hypnotic medication alone or both. Hypnotic medication will include sedating antihistamines, benzodiazepines and non-benzodiazepine hypnotics such as zopiclone. Medication prescribed for dual purpose will be assumed to be used for the treatment of insomnia if given after 2300 hours. Each patient will be enrolled for a period of 4 weeks and the review of use and suitability will take place in ward review meetings.

Sleep quality will be assessed using the Pittsburgh Sleep Quality Assessment tool at baseline and at the 2 and 4 weeks. At the end of the study period, percentage use of amber glasses and zopiclone will be used to compare against a historical average of hypnotic use for the most recent 15 admissions over a similar 4 week period.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Male or female gender
* Presentation of mental illness (of psychotic nature, severe depression or anxiety)
* Able to provide informed consent

Exclusion Criteria:

* Patient does not consent
* High risk assessment of self-harm or harm to others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The difference in the use of hypnotic medication as compared with existing data from a similar population. | 4 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Assessment (PSQI) tool at baseline and at the 2 and 4 weeks. At the end of the study period, percentage use of amber glasses and zopiclone will be used to compare against a historical average of hypnotic use for the most recent 15 admissions over a similar 4 week period. These historic admissions will be matched for diagnosis.

SECONDARY OUTCOMES:
Change in sleep quality as measured by a point score change in the PSQI. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Surrey and Borders NHS Foundation Trust, Leatherhead, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No